CLINICAL TRIAL: NCT05116241
Title: Phase 2b Placebo-Controlled Randomized Study of BPZE1 Intranasal Pertussis Vaccine in Healthy School-Age Children to Assess Immunological Response and Safety of a Single Dose BPZE1 With/Without Coadministration of Tdap (Boostrix™)
Brief Title: Immunogenicity and Safety of BPZE1 Intranasal Pertussis Vaccine in Healthy School-age Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ILiAD Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IB-201P
Record Dates: First submitted 2021-10-20; First posted 2021-11-10 (Actual); Results first posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Bordetella Pertussis, Whooping Cough
Keywords: Bordetella pertussis (B. pertussis); Whooping Cough; BPZE1; Boostrix; Vaccine; Children; Booster; Live attenuated vaccine
MeSH Terms: conditions — Whooping Cough | interventions — Boostrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BPZE1 intranasal and Placebo intramuscular (Experimental): Individual will receive an intranasal dose of BPZE1 via the mucosal atomization device and a dose of intramuscular placebo.
  Interventions: Biological: BPZE1 pertussis vaccine and placebo
- BPZE1 intranasal and Boostrix intramuscular (Experimental): Individual will receive an intranasal dose of BPZE1 via the mucosal atomization device and a dose of intramuscular Boostrix (acellular pertussis [aP] vaccine).
  Interventions: Biological: BPZE1 pertussis vaccine and Boostrix
- Placebo intranasal and Boostrix intramuscular (Active Comparator): Individual will receive an intranasal dose of placebo via the mucosal atomization device and a dose of intramuscular Boostrix (aP vaccine comparator).
  Interventions: Biological: Placebo and Boostrix

INTERVENTIONS:
Biological: BPZE1 pertussis vaccine and placebo — Live attenuated pertussis vaccine and placebo
  Arms: BPZE1 intranasal and Placebo intramuscular
Biological: BPZE1 pertussis vaccine and Boostrix — Live attenuated pertussis vaccine and tetanus, diphtheria, and aP vaccine
  Arms: BPZE1 intranasal and Boostrix intramuscular
Biological: Placebo and Boostrix — Tetanus, diphtheria, and aP vaccine and placebo
  Arms: Placebo intranasal and Boostrix intramuscular

SUMMARY:
This study evaluates the safety and immunogenicity of the BPZE1 live, attenuated pertussis vaccine, intended to prevent nasopharyngeal colonization and pertussis disease, and compares BPZE1 vaccine vs Boostrix vaccine vs both BPZE1 and Boostrix vaccines. This is a multi-center, randomized, placebo- and active-comparator-controlled study in healthy, school-age children with a 6-month safety follow-up after the first vaccination.

DETAILED DESCRIPTION:
This multi-center, randomized, placebo- and active-comparator-controlled study evaluates the safety and immunogenicity of the BPZE1 live attenuated pertussis vaccine, intended to prevent nasopharyngeal colonization and pertussis disease. Healthy school-age children will be randomly assigned to 1 of 3 different study treatment groups to receive the intranasal BPZE1 vaccine, the intramuscular Boostrix vaccine, or both. Subjects will first receive the intranasal vaccine (BPZE1 or placebo) using a small, cone-shaped device that attaches to a syringe and sprays the vaccine into the nose. After a 10-minute waiting period, subjects will receive the intramuscular vaccine (Boostrix or placebo) in the upper arm. As this is the first study in school-age children, a staggered enrollment is planned with the first 45 subjects in the older age group of 11-17 years designated as the safety lead-in cohort. After reactogenicity results from the first 7 days after vaccination of the safety lead-in cohort are reviewed by the safety monitoring committee, the remainder of the subjects will be enrolled. Subjects who choose to take part in a small sub-study of revaccination/attenuated challenge will receive BPZE1 intranasal vaccine (open-label) 3 months after the first vaccination. Safety will be monitored for 6 months after the first vaccination.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female subject 6 to 17 years of age on Day 1.
2. Subject must provide informed consent (assent, depending on age) prior to participation in study and comply with protocol requirements.
3. If female, the subject is not pregnant or lactating. If female of childbearing potential, the subject must agree to either be heterosexually inactive or follow birth control methods per protocol from at least 21 days prior to enrollment and through 90 days following any study vaccination.
4. Subject has a stable health status, as established by physical examination, vital sign measurements, and medical history.
5. Subject (and/or legal guardian) has access to a consistent and reliable means of electronic or telephone contact, which may be in the home, workplace, school, or by personal mobile electronic device.
6. Subject is willing to refrain from routine nasal sprays (including steroid sprays) or washes for at least 7 days following any study vaccination.

Key Exclusion Criteria:

1. The subject has a history of whole-cell pertussis vaccination in lifetime, acellular pertussis-containing vaccination (inclusive of school vaccination programs) within 3 years prior to Day 1, documented B. pertussis infection within 3 years prior to Day 1, or a history of Td-containing vaccination (without pertussis vaccine component) within 1 month prior to Day 1.
2. Chronic significant illness actively being treated or a history of recent intervention for worsening or fluctuating symptoms (at the discretion of the investigator).
3. History of cancer (malignancy).
4. Congenital, hereditary, or acquired disease or disorder classified as autoimmune, immunodeficient, coagulopathy, hepatic, renal, neurologic, or cognitive.
5. Currently uses smoking products (including vaping and e-cigarettes) and is unwilling to refrain from use from Day 1 through Day 29 following study vaccination.
6. Subject received immunoglobulin, blood-derived products, systemic corticosteroids (at a dose of >10 mg per day for more than 10 days), or other immunosuppressant drugs within 90 days of Day 1.
7. Chronic pulmonary disease requiring active medication or pulmonary therapies except exercise-induced bronchospasm, if currently well controlled, and willing to refrain from intense exercise for 7 days following study vaccination, or intermittent asthma classification who have not had an exacerbation requiring oral systemic corticosteroids in the past year; have an forced expiratory volume (FEV1) documented to be >80%; do not have restrictions in normal activity due to breathing issues; and have used a short-acting beta-agonist less than or equal to 2 days per week over the past 2 months.
8. History of oro/nasopharynx surgery (eg, adenoidectomy, tonsillectomy) within 60 days prior to Day 1.
9. Known hypersensitivity to latex or any component of any study vaccine. Specific to Boostrix: hypersensitivity to neomycin or polymyxin; hypersensitivity after previous administration of diphtheria, tetanus, or pertussis vaccines; or has experienced transient thrombocytopenia or neurological complications following an earlier immunization against diphtheria and/or tetanus.
10. Subject has routine and/or repeated contact with, or is currently living in a household with, an immunocompromised individual.
11. Subject resides in a residence where an infant less than 6 months of age resides or may reside.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 368 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- Australia (5):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Sydney Children's Hospital, Westmead, New South Wales
  - Women's and Children's Hospital, North Adelaide, South Australia
  - University of Melbourne, Melbourne, Victoria
  - Telethon Kids Institute, Nedlands, Western Australia
- Costa Rica (3):
  - CSA Clinica San Augustin, San José
  - IICIMED Instituto de Investigacion en Ciencias Medicas, San José
  - MRI, Metropolitan Research Institute, San José
- United Kingdom (8):
  - Birmingham Children's Hospital NHS Foundation Trust, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Bristol Royal Hospital For Children, Bristol
  - Addenbrooke's Hospital, Cambridge
  - Leicester Children's Hospital, Ward 14, Level 4,, Leicester
  - St George's Healthcare NHS Trust, London
  - Oxford Vaccine Group, Oxford
  - University Hospital Southampton NHS Foundation Trust, Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 381 participants screened; 368 participants randomized (2 participants randomized but not vaccinated); 366 participants vaccinated.
  Participants were grouped by age: 6-10 years and 11-17 years with a Safety Lead-in group of 45 participants in the older age group.
  All participants were in the study from 11-Nov-2021 through 15-May-2024
  Period 1 (Day 1): Vaccination; Period 2 (Day 85): Optional Attenuated Challenge Substudy
Groups:
- BPZE1 and Intramuscular Placebo: Day 1: Participants received an intranasal dose of BPZE1 via the mucosal atomization device and a dose of intramuscular placebo.
- BPZE1 and Boostrix Intramuscular: Day 1: Participants received an intranasal dose of BPZE1 via the mucosal atomization device and a dose of intramuscular Boostrix (acellular pertussis [aP] vaccine).
- Placebo Intranasal and Boostrix Intramuscular: Day 1: Participants received an intranasal dose of placebo via the mucosal atomization device and a dose of intramuscular Boostrix (aP vaccine comparator).
Period: Study
Arm/Group | BPZE1 and Intramuscular Placebo | BPZE1 and Boostrix Intramuscular | Placebo Intranasal and Boostrix Intramuscular
Started | 123 | 121 | 122
Completed | 118 | 117 | 119
Not Completed | 5 | 4 | 3
Not completed — Withdrawal by Subject | 5 | 2 | 1
Not completed — Lost to Follow-up | 0 | 2 | 2
Period: Optional Attenuated Challenge Substudy
Arm/Group | BPZE1 and Intramuscular Placebo | BPZE1 and Boostrix Intramuscular | Placebo Intranasal and Boostrix Intramuscular
Started (Enrollment in open-label BPZE1 Attenuated Challenge Substudy (Day 85) was optional and limited to 120 participants.) | 38 | 36 | 46
Completed | 38 | 36 | 46
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- BPZE1 and Intramuscular Placebo: Participants received an intranasal dose of BPZE1 via the mucosal atomization device and a dose of intramuscular placebo.
- BPZE1 and Boostrix Intramuscular: Participants received an intranasal dose of BPZE1 via the mucosal atomization device and a dose of intramuscular Boostrix (acellular pertussis [aP] vaccine).
- Placebo Intranasal and Boostrix Intramuscular: Participants received an intranasal dose of placebo via the mucosal atomization device and a dose of intramuscular Boostrix (aP vaccine comparator).
- Total: Total of all reporting groups
Arm/Group | BPZE1 and Intramuscular Placebo | BPZE1 and Boostrix Intramuscular | Placebo Intranasal and Boostrix Intramuscular | Total
Number analyzed (Participants) | 123 | 121 | 122 | 366
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.9 (2.7) | 10.8 (2.9) | 10.7 (2.8) | 10.8 (2.8)
Age, Customized [Count of Participants; unit: Participants]
  6-10 years | 60 | 67 | 65 | 192
  11-17 years | 63 | 54 | 57 | 174
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 56 | 54 | 170
  Male | 63 | 65 | 68 | 196
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 60 | 58 | 58 | 176
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 63 | 63 | 64 | 190
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 54 | 52 | 55 | 161
  Black | 0 | 0 | 0 | 0
  Asian | 3 | 6 | 0 | 9
  Pacific Islander | 0 | 0 | 0 | 0
  Aboriginal or Torres Strait Islander | 0 | 0 | 0 | 0
  Mixed or Multiple Ethnic Group | 6 | 4 | 10 | 20
  Other Race | 60 | 59 | 57 | 176
Region of Enrollment [Number; unit: participants]
  United Kingdom | 23 | 23 | 22 | 68
  Australia | 27 | 23 | 27 | 77
  Costa Rica | 73 | 75 | 73 | 221

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Mucosal Immunogenicity S-IgA Against Whole Cell Extract at Day 29
Description: Geometric mean fold rise (GMFR) of mucosal S-IgA against whole cell extract (WCE) by treatment arm (BPZE1, BPZE1 + Boostrix) at Day 29.
Time Frame: Day 29
Population: Per protocol immunogenicity analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | BPZE1 and Intramuscular Placebo | BPZE1 and Boostrix Intramuscular | Placebo Intranasal and Boostrix Intramuscular
Number analyzed (Participants) | 105 | 113 | 111
Fold Rise | 3.8 [3.1 to 4.7] | 3.5 [2.9 to 4.3] | 1.2 [1.0 to 1.5]

2. Primary Outcome: Safety: Solicited Adverse Events (AEs)
Description: Solicited AEs (local injection site, nasal/respiratory, and systemic reactogenicity events)
Time Frame: Through 7 days following first study vaccination.
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 and Intramuscular Placebo | BPZE1 and Boostrix Intramuscular | Placebo Intranasal and Boostrix Intramuscular
Number analyzed (Participants) | 123 | 121 | 122
Participants
  Local injection site reactogenicity | 59 | 81 | 88
  Nasal/Respiratory reactogenicity | 61 | 63 | 55
  Systemic reactogenicity | 51 | 60 | 67

3. Secondary Outcome: Serum IgG: Proportion of Subjects With Antibody Concentration ≥0.1 Immunogenicity Serum IgG for Diphtheria, Tetanus
Description: Serum IgG levels against diphtheria, tetanus by treatment groups (BPZE1 + Boostrix vs Boostrix)
Time Frame: Day 29
Population: Per protocol immunogenicity analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 and Boostrix Intramuscular | Placebo Intranasal and Boostrix Intramuscular
Number analyzed (Participants) | 111 | 109
Participants
  Serum IgG against Diphtheria >= 0.1 IU/ml | 111 | 109
  Serum IgG against Tetanus >= 0.1 IU/ml | 111 | 109

4. Secondary Outcome: Serum IgG: Geometric Mean Concentration (GMC) Against Acellular Pertussis Antigens
Description: Serum IgG levels against acellular pertussis antigens (pertussis toxin [PT], filamentous hemagglutinin [FHA], pertactin [PRN]) by treatment groups (BPZE1 + Boostrix vs Boostrix)
Time Frame: Day 29
Population: Per protocol immunogenicity analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | BPZE1 and Boostrix Intramuscular | Placebo Intranasal and Boostrix Intramuscular
Number analyzed (Participants) | 111 | 109
IU/ml
  Serum IgG against PRN | 116.2 [86.9 to 155.4] | 82.5 [57.2 to 118.9]
  Serum IgG against FHA | 502.9 [443.3 to 570.5] | 458.2 [399.8 to 525.1]
  Serum IgG against PT | 88.1 [76.4 to 101.6] | 84.4 [71.9 to 99.0]

5. Secondary Outcome: Mucosal Immunogenicity S-IgA GMR
Description: Induction of normalized S-IgA against WCE, PT, FHA, PRN, and any additional anti-pertussis mucosal antibodies identified during assay development (fimbriae serotype 2 and 3; FIM 2/3) using GMR
Time Frame: Baseline, Day 29
Population: Per protocol immunogenicity analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: AU/(mg S-IgA)
Arm/Group | BPZE1 and Intramuscular Placebo | BPZE1 and Boostrix Intramuscular | Placebo Intranasal and Boostrix Intramuscular
Number analyzed (Participants) | 105 | 113 | 111
AU/(mg S-IgA)
  Baseline WCE | 27.2 [23.8 to 30.9] | 24.8 [21.8 to 28.2] | 22.4 [19.3 to 26.0]
  Baseline PT | 4.0 [3.6 to 4.6] | 3.8 [3.3 to 4.4] | 3.5 [3.1 to 4.0]
  Baseline PRN | 3.0 [2.6 to 3.6] | 3.3 [2.8 to 3.8] | 2.7 [2.3 to 3.1]
  Baseline FHA | 2.3 [2.0 to 2.7] | 2.3 [1.9 to 2.7] | 2.2 [1.9 to 2.7]
  Baseline FIM 2/3 | 3.0 [2.4 to 3.7] | 2.6 [2.2 to 3.0] | 2.3 [1.9 to 2.8]
  Day 29 WCE | 104.0 [86.2 to 125.5] | 86.3 [72.8 to 102.4] | 27.4 [23.6 to 31.7]
  Day 29 PT | 6.8 [5.8 to 7.8] | 6.5 [5.7 to 7.4] | 4.3 [3.8 to 4.9]
  Day 29 PRN | 11.4 [9.3 to 14.1] | 13.6 [11.1 to 16.7] | 4.0 [3.4 to 4.6]
  Day 29 FHA | 18.6 [14.6 to 23.6] | 15.7 [12.8 to 19.2] | 4.7 [3.9 to 5.7]
  Day 29 FIM 2/3 | 42.4 [30.6 to 58.6] | 26.9 [19.6 to 36.9] | 3.0 [2.5 to 3.7]

6. Secondary Outcome: Mucosal Immunogenicity S-IgA GMFR
Description: Induction of normalized S-IgA against WCE, FHA, PRN, and any additional anti-pertussis mucosal antibodies identified during assay development (FIM 2/3) using GMFR
Time Frame: Day 29
Population: Per protocol immunogenicity analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | BPZE1 and Intramuscular Placebo | BPZE1 and Boostrix Intramuscular | Placebo Intranasal and Boostrix Intramuscular
Number analyzed (Participants) | 105 | 113 | 111
Fold Rise
  Day 29 WCE | 3.8 [3.1 to 4.7] | 3.5 [2.9 to 4.3] | 1.2 [1.0 to 1.5]
  Day 29 PT | 1.7 [1.4 to 1.9] | 1.7 [1.5 to 2.0] | 1.2 [1.1 to 1.4]
  Day 29 PRN | 3.7 [2.9 to 4.7] | 4.2 [3.3 to 5.2] | 1.5 [1.3 to 1.8]
  Day 29 FHA | 8.1 [6.1 to 10.8] | 6.8 [5.4 to 8.7] | 2.1 [1.8 to 2.6]
  Day 29 FIM 2/3 | 14.0 [9.6 to 20.5] | 10.5 [7.5 to 14.7] | 1.3 [1.2 to 1.5]

7. Secondary Outcome: Serum Immunogenicity IgA and IgG GMC
Description: Induction of serum immunity (IgA and IgG) against WCE, pertussis toxin (PT), FHA, PRN, and any additional anti-pertussis antibodies identified during assay development (FIM 2/3) using GMC
Time Frame: Baseline, Day 29
Population: Per protocol immunogenicity analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | BPZE1 and Intramuscular Placebo | BPZE1 and Boostrix Intramuscular | Placebo Intranasal and Boostrix Intramuscular
Number analyzed (Participants) | 106 | 111 | 109
IU/ml
  IgG Baseline WCE | 42.4 [35.1 to 51.3] | 52.5 [43.4 to 63.4] | 51.5 [43.2 to 61.2]
  IgG Baseline PT | 7.8 [6.6 to 9.3] | 8.5 [7.2 to 10.1] | 9.1 [7.5 to 10.9]
  IgG Baseline PRN | 7.6 [5.9 to 9.7] | 8.5 [6.6 to 10.8] | 8.4 [6.6 to 10.7]
  IgG Baseline FHA | 31.3 [26.8 to 36.5] | 42.9 [35.9 to 51.1] | 46.2 [37.3 to 57.2]
  IgG Baseline FIM 2/3 | 14.3 [10.6 to 19.3] | 12.9 [10.0 to 16.8] | 13.3 [10.0 to 17.9]
  IgG Day 29 WCE | 111.4 [93.4 to 132.9] | 229.2 [196.0 to 267.9] | 164.9 [142.9 to 190.1]
  IgG Day 29 PT | 31.3 [24.8 to 39.6] | 88.1 [76.4 to 101.6] | 84.4 [71.9 to 99.0]
  IgG Day 29 PRN | 29.3 [23.5 to 36.6] | 116.2 [86.9 to 155.4] | 82.5 [57.2 to 118.9]
  IgG Day 29 FHA | 130.8 [107.3 to 159.4] | 502.9 [443.3 to 570.5] | 458.2 [399.8 to 525.1]
  IgG Day 29 FIM 2/3 | 107.1 [80.8 to 141.8] | 80.2 [61.7 to 104.4] | 21.5 [15.5 to 29.8]
  IgA Baseline WCE | 12.3 [10.9 to 13.8] | 14.7 [12.7 to 17.0] | 14.7 [12.4 to 17.4]
  IgA Baseline PT | 1.5 [1.3 to 1.6] | 1.6 [1.4 to 1.8] | 1.7 [1.4 to 2.0]
  IgA Baseline PRN | 1.5 [1.3 to 1.8] | 1.9 [1.5 to 2.3] | 1.7 [1.4 to 2.2]
  IgA Baseline FHA | 2.2 [1.8 to 2.7] | 2.8 [2.2 to 3.5] | 3.3 [2.5 to 4.3]
  IgA Baseline FIM 2/3 | 2.9 [2.3 to 3.7] | 2.9 [2.3 to 3.6] | 3.3 [2.6 to 4.2]
  IgA Day 29 WCE | 53.0 [44.0 to 63.8] | 56.6 [47.3 to 67.6] | 25.7 [21.3 to 31.1]
  IgA Day 29 PT | 4.3 [3.5 to 5.3] | 4.4 [3.7 to 5.2] | 2.6 [2.2 to 3.0]
  IgA Day 29 PRN | 10.8 [8.4 to 13.8] | 25.0 [18.6 to 33.5] | 6.9 [5.0 to 9.6]
  IgA Day 29 FHA | 20.0 [15.6 to 25.7] | 33.6 [27.3 to 41.3] | 21.1 [16.6 to 27.0]
  IgA Day 29 FIM 2/3 | 45.2 [33.0 to 61.7] | 31.1 [22.2 to 43.7] | 4.5 [3.4 to 6.0]

8. Secondary Outcome: Serum Immunogenicity IgA and IgG GMFR
Description: Induction of serum immunity (IgA and IgG) against WCE, pertussis toxin (PT), FHA, PRN, and any additional anti-pertussis antibodies identified during assay development (FIM 2/3) using GMFR
Time Frame: Baseline, Day 29
Population: Per protocol immunogenicity analysis set
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | BPZE1 and Intramuscular Placebo | BPZE1 and Boostrix Intramuscular | Placebo Intranasal and Boostrix Intramuscular
Number analyzed (Participants) | 106 | 111 | 109
Fold Rise
  IgG Day 29 WCE | 2.6 [2.2 to 3.0] | 4.4 [3.8 to 5.2] | 3.3 [2.8 to 3.8]
  IgG Day 29 PT | 4.0 [3.1 to 5.1] | 10.4 [9.2 to 11.8] | 9.3 [7.8 to 10.9]
  IgG Day 29 PRN | 3.8 [3.0 to 4.8] | 14.5 [11.3 to 18.6] | 9.6 [7.4 to 12.4]
  IgG Day 29 FHA | 4.2 [3.3 to 5.3] | 11.9 [10.0 to 14.3] | 9.9 [8.1 to 12.2]
  IgG Day 29 FIM 2/3 | 7.4 [5.6 to 9.9] | 6.4 [4.9 to 8.3] | 1.7 [1.4 to 1.9]
  IgA Day 29 WCE | 4.2 [3.5 to 5.2] | 3.9 [3.3 to 4.7] | 1.7 [1.5 to 2.1]
  IgA Day 29 PT | 2.9 [2.4 to 3.6] | 2.7 [2.4 to 3.1] | 1.6 [1.4 to 1.8]
  IgA Day 29 PRN | 6.7 [5.4 to 9.1] | 13.9 [10.8 to 17.8] | 4.1 [3.2 to 5.2]
  IgA Day 29 FHA | 9.0 [6.7 to 11.9] | 12.3 [10.0 to 15.1] | 6.7 [5.2 to 8.5]
  IgA Day 29 FIM 2/3 | 15.4 [11.1 to 21.4] | 10.9 [7.7 to 15.3] | 1.4 [1.2 to 1.6]

9. Secondary Outcome: Safety: Reactogenicity and AEs
Description: To describe reactogenicity events during the 7 days following any study vaccination (7 days after Day 1 study vaccination and 7 days after Day 85 attenuated challenge with open-label BPZE1), all AEs through 28 days following Day 1 study vaccination and Day 85 attenuated challenge with open-label BPZE1, medically-attended AEs (MAAE) through 84 days following Day 1 study vaccination and Day 85 attenuated challenge with open-label BPZE1, AEs of special interest (AESIs) and serious adverse events (SAE) through Day 169 (EOS).
Time Frame: Through 7 days, 28 days, and 169 days (EOS) following any study vaccination respectively
Population: Safety Analysis Set for Day 1 includes all vaccinated participants. Safety Analysis Set for Day 85 includes all Attenuated Challenge Open-label BPZE1 Substudy participants.
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 and Intramuscular Placebo | BPZE1 and Boostrix Intramuscular | Placebo Intranasal and Boostrix Intramuscular
Number analyzed (Participants) | 123 | 121 | 122
Participants
  Reactogenicity after Day 1 study vaccination : Local injection site | 59 | 81 | 88
  Reactogenicity after Day 1 study vaccination : Nasal/Respiratory | 61 | 63 | 55
  Reactogenicity after Day 1 study vaccination : Systemic | 51 | 60 | 67
  Reactogenicity after Day 85 attenuated challenge with open-label BPZE1 : Nasal/Respiratory: number analyzed (Participants) | 38 | 36 | 46
  Reactogenicity after Day 85 attenuated challenge with open-label BPZE1 : Nasal/Respiratory | 19 | 16 | 24
  Reactogenicity after Day 85 attenuated challenge with open-label BPZE1 : Systemic: number analyzed (Participants) | 38 | 36 | 46
  Reactogenicity after Day 85 attenuated challenge with open-label BPZE1 : Systemic | 19 | 14 | 22
  Day 29 AEs | 31 | 19 | 26
  Day 85 AEs: number analyzed (Participants) | 38 | 36 | 46
  Day 85 AEs | 4 | 10 | 10
  MAAEs | 25 | 12 | 23
  SAEs | 1 | 0 | 2
  AESI | 4 | 6 | 3

10. Secondary Outcome: Colonization (Substudy Only)
Description: Proportion of subjects with positive B. pertussis by culture or polymerase chain reaction [PCR]) following re-vaccination/attenuated challenge (BPZE1, BPZE1 + Boostrix, BPZE1 and BPZE1 + Boostrix, Boostrix control)
Time Frame: Day 92 or Day 99.
Population: Investigational quantitative PCR not sensitive, no cultures performed and no results available.
Arm/Group | BPZE1 and Intramuscular Placebo | BPZE1 and Boostrix Intramuscular | Placebo Intranasal and Boostrix Intramuscular
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs and deaths collected through end of study - up to 6 months. Unsolicited AEs collected up to 28 days post-vaccination (All participants) and 28 days post-challenge (Only optional Substudy participants).
Groups:
- BPZE1 and Intramuscular Placebo (All Participants Post-vaccination): Participants received an intranasal dose of BPZE1 via the mucosal atomization device and a dose of intramuscular placebo (including all participants, those who participated in the optional substudy and those who did not participate in the optional substudy).
- BPZE1 and Boostrix Intramuscular (All Participants Post-vaccination): Participants received an intranasal dose of BPZE1 via the mucosal atomization device and a dose of intramuscular Boostrix (acellular pertussis [aP] vaccine) (including all participants, those who participated in the optional substudy and those who did not participate in the optional substudy).
- Placebo Intranasal and Boostrix Intramuscular (All Participants Post-vaccination): Participants received an intranasal dose of placebo via the mucosal atomization device and a dose of intramuscular Boostrix (aP vaccine comparator) (including all participants, those who participated in the optional substudy and those who did not participate in the optional substudy).
- BPZE1 and Intramuscular Placebo (Optional Sub-study Participants Post-challenge): Participants received an intranasal dose of BPZE1 via the mucosal atomization device and a dose of intramuscular placebo and also volunteered for the optional substudy.
- BPZE1 and Boostrix Intramuscular (Optional Sub-study Participants Post-challenge): Participants received an intranasal dose of BPZE1 via the mucosal atomization device and a dose of intramuscular Boostrix (acellular pertussis [aP] vaccine) and also volunteered for the optional substudy.
- Placebo Intranasal and Boostrix Intramuscular (Optional Sub-study Participants Post-challenge): Participants received an intranasal dose of placebo via the mucosal atomization device and a dose of intramuscular Boostrix (aP vaccine comparator) and also volunteered for the optional substudy.
Arm/Group | BPZE1 and Intramuscular Placebo (All Participants Post-vaccination) | BPZE1 and Boostrix Intramuscular (All Participants Post-vaccination) | Placebo Intranasal and Boostrix Intramuscular (All Participants Post-vaccination) | BPZE1 and Intramuscular Placebo (Optional Sub-study Participants Post-challenge) | BPZE1 and Boostrix Intramuscular (Optional Sub-study Participants Post-challenge) | Placebo Intranasal and Boostrix Intramuscular (Optional Sub-study Participants Post-challenge)
All-Cause Mortality (participants affected / at risk) | 0/123 | 0/121 | 0/122 | 0/38 | 0/36 | 0/46
Serious Adverse Events (participants affected / at risk) | 1/123 | 0/121 | 2/122 | 0/38 | 0/36 | 0/46
Other Adverse Events (participants affected / at risk) | 31/123 | 19/121 | 26/122 | 4/38 | 10/36 | 10/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BPZE1 and Intramuscular Placebo (All Participants Post-vaccination) (N=123) | BPZE1 and Boostrix Intramuscular (All Participants Post-vaccination) (N=121) | Placebo Intranasal and Boostrix Intramuscular (All Participants Post-vaccination) (N=122) | BPZE1 and Intramuscular Placebo (Optional Sub-study Participants Post-challenge) (N=38) | BPZE1 and Boostrix Intramuscular (Optional Sub-study Participants Post-challenge) (N=36) | Placebo Intranasal and Boostrix Intramuscular (Optional Sub-study Participants Post-challenge) (N=46)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccination. This SAE occurred and resolved prior to optional Sub-study. Participant did volunteer for the optional Sub-study.
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccination. Participant did not volunteer for the optional Sub-study.
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Not related to vaccination. Participant did not volunteer for the optional Sub-study.
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BPZE1 and Intramuscular Placebo (All Participants Post-vaccination) (N=123) | BPZE1 and Boostrix Intramuscular (All Participants Post-vaccination) (N=121) | Placebo Intranasal and Boostrix Intramuscular (All Participants Post-vaccination) (N=122) | BPZE1 and Intramuscular Placebo (Optional Sub-study Participants Post-challenge) (N=38) | BPZE1 and Boostrix Intramuscular (Optional Sub-study Participants Post-challenge) (N=36) | Placebo Intranasal and Boostrix Intramuscular (Optional Sub-study Participants Post-challenge) (N=46)
Upper Respiratory Tract Infection (Infections and infestations) | 7 | 2 | 3 | 0 | 2 | 2 — Day 1 study vaccination
Nasopharyngitis (Infections and infestations) | 2 | 2 | 3 | 0 | 2 | 1 — Day 1 study vaccination
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3 | 1 | 1 | 0 — Day 1 study vaccination
Other (General disorders) | 18 | 14 | 16 | 1 | 5 | 7 — Day 1 study vaccination
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 — Gastroenteritis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/41/NCT05116241/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT05116241/SAP_001.pdf